CLINICAL TRIAL: NCT06037993
Title: Endocannabinoid Activity Remodulation for Psychosis Liability in Youth (EARLY)
Brief Title: Endocannabinoid Activity Remodulation for Psychosis Liability in Youth
Acronym: EARLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Udine (Other)
Collaborators: National Research Council (CNR), Institute of Biomolecular Chemistry (ICB), Italy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-DAME 93/2023
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Clinical High Risk for Psychosis; Ultra High Risk for Psychosis; Attenuated Psychotic Symptoms
Keywords: At-Risk Mental State; Schizophrenia; Endocannabinoid System; Gut-Brain Axis; Palmitoylethanolamide; Nutraceuticals; Prevention; Early Intervention
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: We will evaluate the study viability through an internal pilot that will assess the ability of the study to identify, consent, and follow up CHR patients experiencing APS in the study. We propose a 12-week, open-label, investigator-initiated proof of concept study (Phase-2 Pilot Study) of PEA (600 mg/day) for the treatment of APS in CHR patients. We plan to enrol 20 CHR young adults. Those completing the 12-week initial phase, will be proposed to enter a 24-week extension phase to evaluate the clinical stability of treatment, with the possibility of PEA titration to 1200 mg/day based on clinical improvement obtained so far.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEA arm (Experimental): Palmitoylethanolamide (PEA)-treated patients
  Interventions: Dietary Supplement: Ultra-micronized Palmitoylethanolamide (PEA)

INTERVENTIONS:
Dietary Supplement: Ultra-micronized Palmitoylethanolamide (PEA) — Palmitoylethanolamide (PEA) is an N-acylethanolamine (AE), produced "on demand" by different cell types as a response to actual or potential damage, proven to down-regulate central and peripheral activity of mast cells and non-neuronal cells (e.g., astrocytes, microglia) and to exert protective functions against glutamate neuro-toxicity, accounting for its naturally-occurring anti-inflammatory, analgesic, and anticonvulsant properties. Due to the shared pharmacodynamic properties, PEA is considered as the endogenous equivalent of Cannabidiol (CBD). A growing body of literature has confirmed the role of PEA in most neurobiological mechanisms underpinning several neuropsychiatric conditions both in clinical and preclinical settings. The effect of PEA over neuroinflammation and glutamate signaling may represent a promising biobehavioral mechanism underlying the clinical utility of its oral supplementation in CHR state.

SUMMARY:
Clinical High-Risk (CHR) for Psychosis is characterized by the occurrence of unusual stressful experiences (attenuated psychotic symptoms, APS), anxious symptoms, psychological distress, and substantial impairment of the subject's daily functioning.

It is estimated to be associated with up to 30-35% risk of evolution to frank psychotic disorder within 2-2.5 years. To date, no psychotherapeutic or pharmacological approaches have shown therapeutic evidence in this group of patients.

The aim of this study is to provide a response to an unmet clinical need in this framework of psychic vulnerability by initiating oral therapy with palmitoylethanolamide (PEA), a nutraceutical/food supplement with proven anti-inflammatory and neuroprotective properties.

Indeed, many conditions of psychological distress are thought to be underpinned by systemic inflammatory and/or neuroinflammatory processes, on which PEA has shown remarkable efficacy, including through modulation of the immune response and the interaction between the endocannabinoid system and the gut-microbiota-brain axis.

The trial we are proposing is a 12-week open-label phase 2 study involving the daily intake of PEA 600 mg, at a dosage of 1 tablet/day.

This study will be conducted at the Unit of Psychiatry of Santa Maria della Misericordia Udine University Hospital.

Through this study, we wish to evaluate: the ability of PEA to alleviate APS, anxiety, and psychic distress in CHR-APS individuals; the safety and tolerability of sustained intake of PEA in CHR-APS individuals; and the biological basis of PEA functioning.

The study involves taking PEA orally once daily (600 mg daily) at the same time as a meal during the initial 12-week phase. Upon completion of the initial phase, subjects will be offered to enter an extension phase of the trial of an additional 24 weeks to assess treatment stability, with the possibility of titration of PEA to 1200 mg daily based on observed clinical compensation. Each participant will be on PEA treatment for up to 36 weeks.

During the course of the study, periodic clinical re-evaluations will be conducted at our Day-Hospital setting.

The trial will unfold through one screening visit, one baseline visit, and two follow-up visits (FUP, 4 weeks and 12 weeks apart). The patient will be administered standardized interviews by a qualified investigating physician; clinical objective examination, collection of blood and urine samples for standard hematochemical investigations, collection of blood and stool samples for analysis of some biological markers of interest, monitoring of adherence to therapy intake, side effects, and adverse effects will also be performed during the follow-up visits. The nutraceutical PEA will be dispensed by the clinical investigators at each follow-up visit.

DETAILED DESCRIPTION:
1. STATE OF THE ART Among clinical high-risk (CHR) for psychosis individuals, 30-35 % will develop a full-blown disorder after 2-2.5 years. To date there are no proper tools to predict whoever will evolve to full-blown psychosis nor first-choice interventions to prevent the risk of progression at 6-12 months. The endocannabinoid (eCB) system stands as a mediator of the dopaminergic and glutamatergic systems via the cannabinoid receptor 1 (CB1) in the central nervous system (CNS) and seems to be early altered in psychosis. Cannabidiol (CBD) has shown promising results as a treatment for both psychosis and CHR, especially by regulating eCBs levels via the peroxisome proliferator activated receptors (PPARs). Recent research has focused on the role of eCB-like compounds interacting with non-CB receptors, to identify novel putative pharmacological targets. To this extent, oral palmitoylethanolamide (PEA) supplementation has shown promising therapeutic effects as an adjunctive treatment for patients with schizophrenia negative symptoms and acute mania. Interestingly, PEA peripheral blood levels are elevated in CHR individuals and schizophrenia patients. Oral PEA has shown well-documented safety and tolerability in numerous clinical trials with doses 300-1200 mg per day both in healthy and sick populations. Its nature as an endogenous autacoid and essential human diet compound renders PEA nearly devoid of known or potential adverse effects.
2. DETAILED DESCRIPTION OF THE PROJECT 2.1. RATIONALE FOR CURRENT STUDY

   The main purpose of the present study is to address the absence of an effective treatment for CHR individuals. We will perform an investigator-initiated proof-of-concept study (Phase-2 Pilot Study), with the purpose to examine:

   (i) PEA ability to alleviate subtle psychotic and anxiety symptoms in CHR patients; (ii) PEA safety and tolerability; (iii) The biological basis of PEA effect. 2.2. TRIAL OBJECTIVES

   To evaluate:

   (i) The viability of identifying and consenting CHR patients into a trial with PEA; (ii) The efficacy of PEA in providing relief to attenuated psychotic symptoms (APS) in CHR patients; (iii) Whether sustained PEA treatment is well tolerated by CHR patients over a period of at least 12 weeks; (iv) The biological mechanisms underpinning PEA beneficial effects in CHR patients (e.g., modulation of the endocannabinoid (eCB) system, immunological response, metabolic fingerprinting, gut microbiome composition).

   - Objective (i)

   Feasibility questions:

   Over the first 12 months from first patient recruited we will assess whether:

   (i) A minimum of 20 eligible patients have consented to be enrolled into the study; (ii) At least 80% of recruited patients have completed the 12-week follow-up;

   Feasibility endpoints:

   (i) Number of subjects giving consent; (ii) Proportion of participants completing the 12-week follow-up.

   - Objective (ii)

   Research Questions:

   Our primary clinical research question is whether PEA added to treatment as usual in CHR patients:

   (i) Improves APS;

   Our secondary clinical research questions are whether PEA added to treatment as usual (TAU) in CHR patients:

   (ii) Improves APS to the extent that patients no longer satisfy the diagnostic criteria for CHR; (iii) Relieves the distress associated with APS; (iv) Improves anxiety symptoms; (v) Improves social and role functioning. All the study endpoints for the 12-week clinical trial will be assessed by comparing follow-up (FUP) visits and baseline. For those participants continuing in the 24-week extension phase, change (FUP visit minus baseline) in the severity of psychotic symptoms as measured using the Comprehensive Assessment of At-Risk Mental State (CAARMS) will be compared with the group of those willing to discontinue PEA.
   * Objective (iii) Safety questions: We will evaluate if sustained PEA treatment is well tolerated, with minimal side-effects.

   2.3. PARTICIPANTS

   - Selection of participants: The proposed study will involve a university clinical research facility in Italy. Participants will be enrolled into the internal pilot, that will progress to the open-label trial. Patients who express an interest in the study and are identified as having CHR with APS by their clinical teams will be approached by study researchers and given a patient information sheet. Those who agree to take part in the study will be invited for a screening visit.

   - Heterogeneity in CHR: Being the present study primarily designed to assess the effect of PEA over the symptoms of CHR state and to support clinical homogeneity, we will focus on the CHR-APS sub-group of patients, who are the most severely symptomatic, excluding the other two groups at the screening stage. CHR-APS patients represent the greatest majority (at least 80%) of CHR patients treated by mental health services.

   2.4. INTERVENTION

   - Trial Medication: Oral Palmitoylethanolamide (PEA; 600 mg per day) in tablet form. PEA will be obtained by a pharmaceutical company operating under good manufacturing practice conditions with appropriate certification. The information presented on the labels for PEA will comply with applicable national and local regulations.

   - Dosing Regimen: PEA is to be taken orally once a day (600 mg per day) around mealtime during the 12-week initial phase of the study. During the 24-week extension phase of the study, the trial medication is to be taken from once a day up to twice a day (600-1200 mg per day), based on clinical judgment of the improvement obtained so far, around mealtime. Each participant will undergo PEA treatment for a maximum of 36 weeks. The information presented on the labels for the PEA will comply with applicable national and local regulations.

   - Medication Risks: Being a food supplement/nutraceutical, PEA can be purchased at pharmacies without a medical prescription. While unknown risks cannot be excluded, serious adverse events including overdose have not been documented.

   - Drug Accountability: Study specific prescriptions can be used for dispensing the study product. The study medication will be prescribed by qualified physicians given this role on the study delegation log. Only people designated by the Principal Investigator (PI) can collect medication. Only PEA supplied for this study can be dispensed against the study specific prescription. Full accountability records will be completed including recording the batch, expiry date, people dispensing/checking the prescription, quantity and date of drug returns, empty packaging. Nothing is destroyed without the authorization from the PI.

   - Storage of study medication: PEA will be stored at room temperature (< 25 °C) and not kept in a refrigerator, in compliance with local regulations. It will be stored in a secure area away from other treatments and clearly marked for this study.

   - Removal of study medication outside of expiry date/at trial conclusion and destruction: The expiry date will always be reported on the study medication. Study medication outside of the expiry date will not be dispensed and will be destroyed, subject to authorization, on an ongoing basis.

   - Withdrawal of Subjects: According to Declaration of Helsinki, all participants will have the right to withdraw from the study at any time without giving any reason, without any prejudice to their future medical care, and will be informed as such before consent. A participant's withdrawal will be discussed in terms of only discontinuing the study treatment and continuing follow-up visits. Should the patient request to completely withdraw from the study, the decision will be respected. Already collected data will be kept and included in the final analysis. The investigator themselves may also withdraw participants for various reasons, including but not limited to the following: protocol violations, inter-current illness, adverse events, serious adverse events, suspected unexpected serious adverse reactions, administrative reasons, participation in the trial affecting their ongoing care, symptomatic worsening. In the latter case, patients will be followed up with the same schedule of research assessments as those who continue in the study, till they complete the 12-week follow-up period or till they progress to frank psychosis (whichever is earlier). In case of CHR patients experiencing progression to a first episode of psychosis, they will exit from the study intervention, be deemed as treatment failure, and will only be assessed for safety outcomes until they complete the 12-week follow-up period.

   - Subject Compliance: Pill-counts will be performed at FUP visits 1, 2, 3, and 4, to assess compliance with PEA treatment. Patients will be defined as complying in the presence of a pill count greater than 50% the expected number taken. Patients who are defined as non-complying with the medication will be coded as protocol deviators.

   - Concomitant Medication: Based on participants' clinical history, concomitant requirement of psychotropic medication is an exclusion criterion for the study, except for patients undergoing Selective Serotonin Reuptake Inhibitor (SSRI) stable monotherapy (at least 8 months). Patients requiring continued treatment with other classes of psychotropic medications during the treatment phase may be withdrawn from the study by the PI. Very short-term treatment with rescue medications that have a well-established sedative or calming effect (e.g., Benzodiazepines) during the study may be allowed. Throughout the study, any other concomitant medications or treatments deemed necessary to provide adequate supportive care may be prescribed by investigators. A record will be kept listing all concomitant medications received during the treatment phase.

   2.5. VISIT ASSESSMENTS

   The following visit assessments will be performed:
   * First Screening Visit: Approximately one week prior to the Second Screening Visit and two to three weeks prior to the Baseline Visit. Informed consent will be obtained from those who wish to take part to the study. Consenting patients will then be screened against the study inclusion and exclusion criteria using the CAARMS and collecting information on their medical history and substance use information. Individuals satisfying the criteria will be recruited by employed or delegated investigators. Also, consent will be obtained on all participants screened to collect plasma/serum/urine/fecal samples for routine biochemistry and hematology, endocannabinoid, immune, metabolic, and gut microbiome analysis. Consent will be sought to analyze screening data as well as regarding long-term follow-up beyond the outcomes of the trial and to link participants' data to routinely collected data sources such as Hospital Episode Statistics and General Practitioner records.
   * Second Screening Visit: One to two weeks prior to Baseline Visit. Safety blood and urine samples (for routine biochemistry and hematology) will be obtained, physical examination and vital signs will be recorded.
   * Baseline Visit (day 0): Following satisfactory completion of screening, baseline measures (CAARMS, HADS, Global Functioning), physical examination, blood, and fecal samples for endocannabinome (eCBome), immune, metabolic, and gut microbiota analyses will be acquired. Patients will be prescribed PEA and the medication will be dispensed. Side effects will also be assessed, by using the UKU side-effect rating scale.
   * FUP Visit 1 (Week 4 ± 7 days, approximately day 28): At Month 1 and involve clinical assessments (CAARMS, HADS, Global Functioning), blood, and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects, adverse events, and dispensing of study drugs.
   * FUP Visit 2 (Week 12 ± 14 days, approximately Day 84): This visit will be carried out at Month 3 and involve clinical measures (CAARMS, HADS, Global Functioning), physical examination, safety blood and urine samples, blood and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects, adverse events, and dispensing of study drugs.
   * FUP Visit 3 (Week 24 ± 14 days, approximately Day 168): This visit will be carried out at Month 6 on those enrolled in the extension phase and involve clinical assessments (CAARMS, HADS, Global Functioning), blood and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects, adverse events, and dispensing of study drugs.
   * FUP Visit 4 (Week 36 ± 14 days, at approximately Day 252): This visit will be carried out at Month 9 on those enrolled in the extension phase and involve clinical measures (CAARMS, HADS, Global Functioning), physical examination, safety blood and urine samples, blood and fecal sampling for eCBome, immune, metabolic, and gut microbiota analyses, monitoring of compliance, side effects, adverse events, and dispensing of study drugs.
   * Laboratory Tests: Blood tests for hematology (Full blood count and Hemoglobin), biochemistry (Urea & Electrolytes, liver function test, lipid profile), and immune profile characterization will be carried out at the clinical research recruitment hub as per their standard procedure. Blood results will be printed and filed as source in the patient folder. Serum samples for performing metabolic fingerprinting by Raman Spectroscopy, as well as blood and fecal samples for measurement of the levels of eCBome mediators and determination of the microbial composition in feces by Next Generation Sequencing (NGS) of 16SRNA and shotgun metagenomics methodologies, will be shipped to counseling specialized centers where they will be stored and analyzed.

   2.6. SAMPLE SIZE - Proposed sample size: We aim at enrolling 20 patients within 12 months from the start of recruitment.

   - Sample size justification: The number is coherent with suggested sample sizes for pilot studies and is deemed sufficient to evaluate feasibility outcomes. No powered sample size calculation was implemented for the pilot study.

   2.7. METHODS

   - Data collection, management and archiving: Assessment and collection of baseline, outcome and other trial data will be performed according to Visit assessments flow-chart. In case of trial intervention discontinuation, follow-up data will be collected anyway, unless a participant expresses the wish to be completely withdrawn from the study. All data source will be held on as a paper source data worksheet (SDW). These will be managed locally under the care of the recruiting and consenting site PI. Collected data will be held on paper SDW which will be thereafter recorded by allowed study team members on a 24-hour-accessible electronic-based data entry system hosted by the clinical research recruitment hub at ASUFC and University of Udine, consenting data entry to run in parallel with participant enrolment and visits. At the conclusion of the trial the study team will have resolved the data queries and request to remove user access to ensure that the final dataset cannot be changed. SDWs, electronic-based data, and the final statistical report will be archived. Systems will be in place to secure the data collection system against permanent loss and allow the recovery and restoration in the event of such a loss occurring.

   - Data verification, statistical monitoring and analysis: At the study start, a structured data verification plan will be agreed and developed by the Head Statistician of the research team. Data will be checked for consistency across paper- and electronic-based entry systems. Statistical monitoring will include patient severity level, eventual withdrawals, baseline data, FUP visits data, and AEs. The research team will approve a Statistical Analysis Plan within the early stages of the study, and before the Head Statistician summarizes any data. Proportions will be presented for each feasibility outcome. Interim analyses are not planned. The Head Statistician will both carry out and interpret statistical analysis. Our primary analysis will involve a generalized linear model with CAARMS psychotic symptom severity as the dependent measure and time as a repeated measure within subject. We are interested in whether there is a significant benefit over time with PEA treatment. CAARMS distress and total score as well as HADS ratings will be analysed in a similar manner. We will also conduct paired t tests based on baseline and endpoint assessments to examine measures of CAARMS severity and secondary measures. Rates of side effects will be reported, as well as reasons for dropouts from the trial.

   - Missing Data: We expect withdrawn patients to be missing at random, and very few participants withdrawing consent. All patients having at least one post-baseline outcome measure, would be included in each analysis. Nonetheless, patterns of missing data will be explored to investigate any evidence against missing at random, whose impact on the analysis will be considered by introducing imputation methods.

   2.8. ETHICS

   - Ethics & Regulatory Approvals: The trial will be conducted in accordance with the principles of the Declaration of Helsinki (1996), the principles of Good Clinical Practice (GCP), and with all applicable regulatory requirements. This protocol and related documents will be submitted for review to the local Research Ethics Committee (REC).

   - Consent Prior to Screening: Those expressing interest into the study will be referred to the clinical research recruitment hub by their consultants. At screening, investigators will introduce the trial and provide the patients with exhaustive Patient Information Sheets (PIS). Allowed qualified physicians will discuss the trial with patients in light of the information provided in the PIS and give appropriate time for the participants to understand the information provided, before asking written informed consent from those willing to take part to the trial.

   - Biological Samples: The collection of routine blood samples, urine samples, fecal samples, and genotyping will be specifically addressed through the collection of ad hoc consent for biological materials. After collection at the research recruitment hub, obtained blood samples for haematology, biochemistry, and Immune profile characterization will be delivered by the study research team to the local laboratory for analysis. Blood and fecal samples collected to perform metabolic fingerprinting, measurement of the levels of eCBome mediators, and determination of the microbial composition, will be stored in local facilities under adequate conditions (-80°C) and then shipped to counseling specialized centers for subsequent analysis.

   2.9. CONFIDENTIALITY All study-related information will be stored securely at the study site. All participant information will be stored in locked file cabinets in areas with limited access. All laboratory specimens, reports, data collection, process, and administrative forms will be identified by a coded identification (ID) number only to maintain participant confidentiality. All records that contain names or other personal identifiers, such as locator forms and informed consent forms, will be stored separately from study records identified by code number. All local databases will be secured with password-protected access systems. Forms, lists, logbooks, appointment books, and any other listings that link participant ID numbers to other identifying information will be stored in a separate, locked file in an area with limited access. Participants' study information will not be released outside of the study without the written permission of the participant.
3. DISSEMINATION POLICY The results of the study are intended to be reported and disseminated at national/international conferences and in peer-reviewed scientific journals. Our objective is to submit for publication the main results of the trial within two years of last patient recruitment.

ELIGIBILITY:
Inclusion Criteria

* Individuals diagnosed with CHR-APS, as defined using CAARMS criteria;
* Aged 18-35 years;
* To be able to understand and communicate in Italian;
* To be able to give informed consent.

Exclusion Criteria

* Lifetime history of a psychotic or manic episode lasting 7 days or longer;
* Active suicidal ideation indicating significant current risk or history of serious suicide attempt in the opinion of the PI, as evaluated at the screening stage;
* Lifetime neurological disorders (e.g., epilepsy, except febrile convulsions) or severe intercurrent physical illness;
* Current treatment with psychotropic medication, with the exception of Selective Serotonin Reuptake Inhibitor (SSRI) stable monotherapy (at least 8 months);
* Lifetime treatment with antipsychotic medication for more than 7 days;
* IQ < 70;
* Female patients who are pregnant, lactating or not using an acceptable effective form contraception if they are at risk of falling pregnant;
* Taking part in another pharmacological trial.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Severity of attenuated psychotic symptoms (APS) | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Comprehensive Assessment of At-Risk Mental State (CAARMS)

SECONDARY OUTCOMES:
Distress associated with psychotic symptoms | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Comprehensive Assessment of At-Risk Mental State (CAARMS)
Severity of anxiety symptoms | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Hospital Anxiety and Depression Scale (HADS)
Level of impaired global functioning | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Social and Role functioning Scale
Clinical remission, defined as no longer meeting the APS criteria | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Comprehensive Assessment of At-Risk Mental State (CAARMS)
Total CAARMS score | 12 weeks for the initial phase, further 24 weeks for the extension phase
  Comprehensive Assessment of At-Risk Mental State (CAARMS)

OTHER OUTCOMES:
Safety endpoints: Incidence of adverse effects during the study period | 12 weeks for initial phase, further 24 weeks for the extension phase
  UKU side-effect rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Marco Colizzi, MD, PhD, Principal Investigator — University of Udine
Locations (2):
- Italy (2):
  - Unit of Psychiatry, University Hospital of Udine, Udine, UD
  - Unit of Psychiatry, University Hospital of Udine, Udine

REFERENCES:
- [Derived] Bortoletto R, Garzitto M, Basaldella M, Scipioni C, Sepulcri O, Fabris M, Curcio F, Balestrieri M, Colizzi M. Effects of palmitoylethanolamide in clinical high-risk for psychosis: A nonrandomized open-label trial. Brain Behav Immun Health. 2025 Nov 22;50:101141. doi: 10.1016/j.bbih.2025.101141. eCollection 2025 Dec. PMID 41378189
- See also: Questioning the role of palmitoylethanolamide in psychosis: a systematic review of clinical and preclinical evidence — https://www.frontiersin.org/articles/10.3389/fpsyt.2023.1231710/full
- See also: Therapeutic effect of palmitoylethanolamide in cognitive decline: A systematic review and preliminary meta-analysis of preclinical and clinical evidence — https://www.frontiersin.org/articles/10.3389/fpsyt.2022.1038122/full
- See also: Cannabidiol enhances anandamide signaling and alleviates psychotic symptoms of schizophrenia — https://www.nature.com/articles/tp201215
- See also: Childhood trauma and being at-risk for psychosis are associated with higher peripheral endocannabinoids — https://www.cambridge.org/core/journals/psychological-medicine/article/abs/childhood-trauma-and-being-atrisk-for-psychosis-are-associated-with-higher-peripheral-endocannabinoids/BFFDA252EF2250C2F2B45786CC152CDC